CLINICAL TRIAL: NCT05942339
Title: Study on Preliminary Safety and Efficacy of the ARC Therapy Using the ARC-IM Lumbar System to Support Mobility in People With Chronic Spinal Cord Injury
Brief Title: Study on Preliminary Safety and Efficacy of the ARC Therapy Using the ARC-IM Lumbar System to Support Mobility in People With Chronic Spinal Cord Injury (BoxSwitch)
Acronym: BoxSwitch
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ecole Polytechnique Fédérale de Lausanne (Other)
Responsible Party: Principal Investigator, Jocelyne Bloch, Professor, Neurosurgeon, Centre Hospitalier Universitaire Vaudois
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BOX2023
Record Dates: First submitted 2023-06-12; First posted 2023-07-12 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Spinal Cord Injuries
Keywords: SCI; Spinal Cord Injury; Epidural Spinal Stimulation
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Single-site, single-arm, non-blinded, non-randomized, interventional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Targeted Epidural Spinal Stimulation (Experimental): Single arm study: the participants who have previously received a spinal array and an implantable pulse generator either through the STIMO study or similar studies conducted abroad will be proposed to exchange their currently implanted system with selected components from the ARC-IM Lumbar system.
  After the surgery, the participants will perform around 20 optimization sessions that may include rehabilitation to configure the neuromodulation system. Then the participants will use the ARC-IM Lumbar system independently during daily life activities until the end of the 36 months post-surgery. Assessments will be planned throughout the course of the study at the end of the optimization phase, after 12 and 24 months post-surgery and at the end of the study, with and/or stimulation.
  Interventions: Device: Procedure/Surgery

INTERVENTIONS:
Device: Procedure/Surgery — The intervention involves the replacement of parts of the current implanted system with components of the ARC-IM Lumbar system.

SUMMARY:
The purpose of this pre-market clinical study is to assess the preliminary safety and efficacy of the ARC Therapy using the ARC-IM Lumbar System at supporting mobility in participants who have previously received a spinal array and an implantable pulse generator (IPG) either through the STIMO protocol (NCT02936453) or similar studies conducted abroad. They will be proposed to exchange their currently implanted system with components of the newly developed ARC-IM Lumbar system. The goal is to improve more effective lower-limb motor activities, while also simplifying the personal at-home use of the system. In addition, this study aims to evaluate the potential effect of ARC Therapy on muscle tone, bladder, bowel and sexual functions, and quality of life of the participants.

Preliminary safety and efficacy will be assessed in both the short term and throughout the duration of the study (from the surgery to 36 months after the implantation of the ARC-IM Lumbar system).

DETAILED DESCRIPTION:
Studies have shown that using Electrical Epidural Stimulation (EES) could improve considerably the functional movements after paralyzing SCI. In the STIMO study (NCT02936453), the investigational system was mainly composed of medical devices developed for other indications and used off-label, allowing only a limited tuning of EES protocols. To overcome this limitation, we propose to conduct a study in which a new platform will be investigated. This new therapy, named ARC Therapy, features the ARC-IM implantable pulse generator with an optimized communication system and the ARC-IM implantable leads supporting stimulation protocols specifically developed for effective activation of motor neurons.

The study will take place at the CHUV (Lausanne, Switzerland). A maximum of 8 participants will be enrolled in the study and implanted with an ARC-IM IPG. Patients who previously received an implantation in international studies for continuous electrical stimulation can enroll in the current BoxSwitch study. Replacement of their currently implanted IPG and lead will be assessed on a case-by-case manner considering current status of their implanted devices, technical and surgical compatibility with the newly proposed ARC-IM Lumbar system components.

The study intervention consists of several phases preceded by pre-screening:

Screening and enrollment, baseline and pre-implantation assessments, surgery, optimization phase, short-term assessments, independent use phase and follow-up assessments at months 12, 24 and 36. Measures will be performed before surgical intervention and at regular intervals during the study.

The total duration of the study will be approximately 48 months (up to 36 months/participant).

ELIGIBILITY:
Inclusion Criteria:

1. Implanted with a spinal array (Specify 5-6-5 or Go2 Lead) for lower limb mobility, as confirmed by imaging, videos, or neurophysiology recordings.
2. Age 18-65
3. SCI graded as American Spinal Injury Association Impairment Scale (AIS) A, B, C & D
4. SCI ≥ 12months
5. SCI lesion level T10 and above with preservation of conus function
6. SCI due to trauma
7. Stable medical, physical and psychological condition as considered by the investigators
8. Able to understand and interact with the study team in French or English
9. Agrees to comply in good faith with all conditions of the study and to attend all scheduled appointments
10. Must provide and sign the Informed Consent prior to any study-related procedures

Exclusion Criteria:

1. Diseases and conditions that would increase the morbidity and mortality of spinal cord injury surgery
2. History of myocardial infarction or cerebrovascular event within the past 6 months
3. Limitation of walking function based on accompanying (CNS) disorders (systemic malignant disorders, cardiovascular disorders restricting physical training, peripheral nerve disorders)
4. Any active implanted cardiac device such as pacemaker or defibrillator
5. Any indication that would require diathermy
6. Any indication that would require MRI
7. Any anatomical limitations in the implantation area as judged by the investigators
8. Other conditions that would make the subject unable to participate in testing in the judgement of the investigators
9. Clinically significant mental illness in the judgement of the investigators
10. Presence of indwelling baclofen or insulin pump
11. Other clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease, etc.)
12. Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, or dementia of the participant
13. Enrolment of the investigator, his/her family members, employees, and other dependent persons
14. Women who are pregnant (pregnancy test obligatory for women of childbearing potential) or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Preliminary safety of the ARC Therapy | Through study completion (expected 3 years)
  Occurrence of Serious Adverse Events and Adverse Events that are deemed related or possibly related to the study procedure or to the ARC-IM system.

SECONDARY OUTCOMES:
10 Meters Walk test (m/s) | Baseline, Short-term (up to 6months), 12 months, 24 months and 36 months
  The 10 Meters Walk Test is a performance measure used to assess walking speed in meters per second over a short distance.
6 Minutes Walk test (meters) | Baseline, Short-term (up to 6months), 12 months, 24 months and 36 months
  The 6 minutes walk test is a performance measureused to assess aerobic capacity and endurance.
International Standards For Neurological Classification of Spinal Injury (ISNCSCI) | Baseline, 12 months, 24 months and 36 months
  A neurological assessment and classification of a spinal cord injury
Spinal Cord Injury Functional Ambulation Inventory (SCI-FAI) | Baseline, Short-term (up to 6months), 12 months, 24 months and 36 months
  The SCI-FAI assesses functional walking ability in ambulatory individuals with SCI.
Neuromuscular Recovery Scale (NRS) | Baseline, Short-term (up to 6months), 12 months, 24 months and 36 months
  The NRS is used to measure quality of movement without compensatory movement patterns using a body weight support system and a treadmill.
Walking Index for Spinal Cord Injury (WISCI II) | Baseline, Short-term (up to 6months), 12 months, 24 months and 36 months
  The Walking Index for Spinal Cord Injury (WISCI) is a scale that measures the type and amount of assistance (in terms of requirements of assistive devices, or human helpers) required by a person with spinal cord injury (SCI) for walking.
Modified Ashworth Scale (MAS) | Baseline, Short-term (up to 6months), 12 months, 24 months and 36 months
  The modified Ashworth scale a universally accepted clinical tool used to measure the increase of muscle tone.
Spinal Cord Independence Measure (SCIM III) | Baseline, Short-term (up to 6months), 12 months, 24 months and 36 months
  The SCIM address specific areas of function in patients with spinal cord injuries (SCI).
Quality of Life questionnaires | Monthly during the first year
  Questionnaires addressing bowel, bladder and sexual functions.

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyne Bloch, MD, Principal Investigator — CHUV
Locations (1):
- CHUV, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anderson KD. Targeting recovery: priorities of the spinal cord-injured population. J Neurotrauma. 2004 Oct;21(10):1371-83. doi: 10.1089/neu.2004.21.1371. PMID 15672628
- [Background] Cragg JJ, Noonan VK, Krassioukov A, Borisoff J. Cardiovascular disease and spinal cord injury: results from a national population health survey. Neurology. 2013 Aug 20;81(8):723-8. doi: 10.1212/WNL.0b013e3182a1aa68. Epub 2013 Jul 24. PMID 23884034
- [Background] West CR, Phillips AA, Squair JW, Williams AM, Walter M, Lam T, Krassioukov AV. Association of Epidural Stimulation With Cardiovascular Function in an Individual With Spinal Cord Injury. JAMA Neurol. 2018 May 1;75(5):630-632. doi: 10.1001/jamaneurol.2017.5055. PMID 29459943
- [Background] Brinkhof MW, Al-Khodairy A, Eriks-Hoogland I, Fekete C, Hinrichs T, Hund-Georgiadis M, Meier S, Scheel-Sailer A, Schubert M, Reinhardt JD; SwiSCI Study Group. Health conditions in people with spinal cord injury: Contemporary evidence from a population-based community survey in Switzerland. J Rehabil Med. 2016 Feb;48(2):197-209. doi: 10.2340/16501977-2039. PMID 26931074
- [Background] Krassioukov A, Eng JJ, Warburton DE, Teasell R; Spinal Cord Injury Rehabilitation Evidence Research Team. A systematic review of the management of orthostatic hypotension after spinal cord injury. Arch Phys Med Rehabil. 2009 May;90(5):876-85. doi: 10.1016/j.apmr.2009.01.009. PMID 19406310
- [Background] Formento E, Minassian K, Wagner F, Mignardot JB, Le Goff-Mignardot CG, Rowald A, Bloch J, Micera S, Capogrosso M, Courtine G. Electrical spinal cord stimulation must preserve proprioception to enable locomotion in humans with spinal cord injury. Nat Neurosci. 2018 Dec;21(12):1728-1741. doi: 10.1038/s41593-018-0262-6. Epub 2018 Oct 31. PMID 30382196
- [Background] Phillips AA, Krassioukov AV. Contemporary Cardiovascular Concerns after Spinal Cord Injury: Mechanisms, Maladaptations, and Management. J Neurotrauma. 2015 Dec 15;32(24):1927-42. doi: 10.1089/neu.2015.3903. Epub 2015 Sep 1. PMID 25962761
- [Background] Kathe C, Skinnider MA, Hutson TH, Regazzi N, Gautier M, Demesmaeker R, Komi S, Ceto S, James ND, Cho N, Baud L, Galan K, Matson KJE, Rowald A, Kim K, Wang R, Minassian K, Prior JO, Asboth L, Barraud Q, Lacour SP, Levine AJ, Wagner F, Bloch J, Squair JW, Courtine G. The neurons that restore walking after paralysis. Nature. 2022 Nov;611(7936):540-547. doi: 10.1038/s41586-022-05385-7. Epub 2022 Nov 9. PMID 36352232
- [Background] Claydon VE, Steeves JD, Krassioukov A. Orthostatic hypotension following spinal cord injury: understanding clinical pathophysiology. Spinal Cord. 2006 Jun;44(6):341-51. doi: 10.1038/sj.sc.3101855. Epub 2005 Nov 22. PMID 16304564
- [Background] Skinnider MA, Squair JW, Kathe C, Anderson MA, Gautier M, Matson KJE, Milano M, Hutson TH, Barraud Q, Phillips AA, Foster LJ, La Manno G, Levine AJ, Courtine G. Cell type prioritization in single-cell data. Nat Biotechnol. 2021 Jan;39(1):30-34. doi: 10.1038/s41587-020-0605-1. Epub 2020 Jul 20. PMID 32690972
- [Background] Squair JW, Skinnider MA, Gautier M, Foster LJ, Courtine G. Prioritization of cell types responsive to biological perturbations in single-cell data with Augur. Nat Protoc. 2021 Aug;16(8):3836-3873. doi: 10.1038/s41596-021-00561-x. Epub 2021 Jun 25. PMID 34172974
- [Background] Squair JW, Gautier M, Kathe C, Anderson MA, James ND, Hutson TH, Hudelle R, Qaiser T, Matson KJE, Barraud Q, Levine AJ, La Manno G, Skinnider MA, Courtine G. Confronting false discoveries in single-cell differential expression. Nat Commun. 2021 Sep 28;12(1):5692. doi: 10.1038/s41467-021-25960-2. PMID 34584091
- [Background] Gill M, Linde M, Fautsch K, Hale R, Lopez C, Veith D, Calvert J, Beck L, Garlanger K, Edgerton R, Sayenko D, Lavrov I, Thoreson A, Grahn P, Zhao K. Epidural Electrical Stimulation of the Lumbosacral Spinal Cord Improves Trunk Stability During Seated Reaching in Two Humans With Severe Thoracic Spinal Cord Injury. Front Syst Neurosci. 2020 Nov 19;14:79. doi: 10.3389/fnsys.2020.569337. eCollection 2020. PMID 33328910
- [Background] Grindberg RV, Yee-Greenbaum JL, McConnell MJ, Novotny M, O'Shaughnessy AL, Lambert GM, Arauzo-Bravo MJ, Lee J, Fishman M, Robbins GE, Lin X, Venepally P, Badger JH, Galbraith DW, Gage FH, Lasken RS. RNA-sequencing from single nuclei. Proc Natl Acad Sci U S A. 2013 Dec 3;110(49):19802-7. doi: 10.1073/pnas.1319700110. Epub 2013 Nov 18. PMID 24248345
- [Background] Lake BB, Ai R, Kaeser GE, Salathia NS, Yung YC, Liu R, Wildberg A, Gao D, Fung HL, Chen S, Vijayaraghavan R, Wong J, Chen A, Sheng X, Kaper F, Shen R, Ronaghi M, Fan JB, Wang W, Chun J, Zhang K. Neuronal subtypes and diversity revealed by single-nucleus RNA sequencing of the human brain. Science. 2016 Jun 24;352(6293):1586-90. doi: 10.1126/science.aaf1204. PMID 27339989
- [Background] Maniatis S, Aijo T, Vickovic S, Braine C, Kang K, Mollbrink A, Fagegaltier D, Andrusivova Z, Saarenpaa S, Saiz-Castro G, Cuevas M, Watters A, Lundeberg J, Bonneau R, Phatnani H. Spatiotemporal dynamics of molecular pathology in amyotrophic lateral sclerosis. Science. 2019 Apr 5;364(6435):89-93. doi: 10.1126/science.aav9776. PMID 30948552
- [Background] Stahl PL, Salmen F, Vickovic S, Lundmark A, Navarro JF, Magnusson J, Giacomello S, Asp M, Westholm JO, Huss M, Mollbrink A, Linnarsson S, Codeluppi S, Borg A, Ponten F, Costea PI, Sahlen P, Mulder J, Bergmann O, Lundeberg J, Frisen J. Visualization and analysis of gene expression in tissue sections by spatial transcriptomics. Science. 2016 Jul 1;353(6294):78-82. doi: 10.1126/science.aaf2403. PMID 27365449
- [Background] Asboth L, Friedli L, Beauparlant J, Martinez-Gonzalez C, Anil S, Rey E, Baud L, Pidpruzhnykova G, Anderson MA, Shkorbatova P, Batti L, Pages S, Kreider J, Schneider BL, Barraud Q, Courtine G. Cortico-reticulo-spinal circuit reorganization enables functional recovery after severe spinal cord contusion. Nat Neurosci. 2018 Apr;21(4):576-588. doi: 10.1038/s41593-018-0093-5. Epub 2018 Mar 19. PMID 29556028
- [Background] Mignardot JB, Le Goff CG, van den Brand R, Capogrosso M, Fumeaux N, Vallery H, Anil S, Lanini J, Fodor I, Eberle G, Ijspeert A, Schurch B, Curt A, Carda S, Bloch J, von Zitzewitz J, Courtine G. A multidirectional gravity-assist algorithm that enhances locomotor control in patients with stroke or spinal cord injury. Sci Transl Med. 2017 Jul 19;9(399):eaah3621. doi: 10.1126/scitranslmed.aah3621. PMID 28724575
- [Background] Wagner FB, Mignardot JB, Le Goff-Mignardot CG, Demesmaeker R, Komi S, Capogrosso M, Rowald A, Seanez I, Caban M, Pirondini E, Vat M, McCracken LA, Heimgartner R, Fodor I, Watrin A, Seguin P, Paoles E, Van Den Keybus K, Eberle G, Schurch B, Pralong E, Becce F, Prior J, Buse N, Buschman R, Neufeld E, Kuster N, Carda S, von Zitzewitz J, Delattre V, Denison T, Lambert H, Minassian K, Bloch J, Courtine G. Targeted neurotechnology restores walking in humans with spinal cord injury. Nature. 2018 Nov;563(7729):65-71. doi: 10.1038/s41586-018-0649-2. Epub 2018 Oct 31. PMID 30382197
- [Background] Phillips AA, Krassioukov AV, Ainslie PN, Warburton DE. Baroreflex function after spinal cord injury. J Neurotrauma. 2012 Oct 10;29(15):2431-45. doi: 10.1089/neu.2012.2507. Epub 2012 Sep 20. PMID 22897489
- [Background] Rowald A, Komi S, Demesmaeker R, Baaklini E, Hernandez-Charpak SD, Paoles E, Montanaro H, Cassara A, Becce F, Lloyd B, Newton T, Ravier J, Kinany N, D'Ercole M, Paley A, Hankov N, Varescon C, McCracken L, Vat M, Caban M, Watrin A, Jacquet C, Bole-Feysot L, Harte C, Lorach H, Galvez A, Tschopp M, Herrmann N, Wacker M, Geernaert L, Fodor I, Radevich V, Van Den Keybus K, Eberle G, Pralong E, Roulet M, Ledoux JB, Fornari E, Mandija S, Mattera L, Martuzzi R, Nazarian B, Benkler S, Callegari S, Greiner N, Fuhrer B, Froeling M, Buse N, Denison T, Buschman R, Wende C, Ganty D, Bakker J, Delattre V, Lambert H, Minassian K, van den Berg CAT, Kavounoudias A, Micera S, Van De Ville D, Barraud Q, Kurt E, Kuster N, Neufeld E, Capogrosso M, Asboth L, Wagner FB, Bloch J, Courtine G. Activity-dependent spinal cord neuromodulation rapidly restores trunk and leg motor functions after complete paralysis. Nat Med. 2022 Feb;28(2):260-271. doi: 10.1038/s41591-021-01663-5. Epub 2022 Feb 7. PMID 35132264
- [Background] Capogrosso M, Wenger N, Raspopovic S, Musienko P, Beauparlant J, Bassi Luciani L, Courtine G, Micera S. A computational model for epidural electrical stimulation of spinal sensorimotor circuits. J Neurosci. 2013 Dec 4;33(49):19326-40. doi: 10.1523/JNEUROSCI.1688-13.2013. PMID 24305828
- [Background] Greiner N, Barra B, Schiavone G, Lorach H, James N, Conti S, Kaeser M, Fallegger F, Borgognon S, Lacour S, Bloch J, Courtine G, Capogrosso M. Recruitment of upper-limb motoneurons with epidural electrical stimulation of the cervical spinal cord. Nat Commun. 2021 Jan 19;12(1):435. doi: 10.1038/s41467-020-20703-1. PMID 33469022
- [Background] Moraud EM, Capogrosso M, Formento E, Wenger N, DiGiovanna J, Courtine G, Micera S. Mechanisms Underlying the Neuromodulation of Spinal Circuits for Correcting Gait and Balance Deficits after Spinal Cord Injury. Neuron. 2016 Feb 17;89(4):814-28. doi: 10.1016/j.neuron.2016.01.009. Epub 2016 Feb 4. PMID 26853304
- [Background] Minassian K, Hofstoetter U, Tansey K, Mayr W. Neuromodulation of lower limb motor control in restorative neurology. Clin Neurol Neurosurg. 2012 Jun;114(5):489-97. doi: 10.1016/j.clineuro.2012.03.013. Epub 2012 Mar 29. PMID 22464657